CLINICAL TRIAL: NCT06812052
Title: Prospective Phase I Trial of Hypofractionated Radiation Therapy in Retroperitoneal Sarcoma
Brief Title: Short Course Radiation Treatment for Patients With Primary or Locally Recurrent Retroperitoneal Sarcoma Prior to Surgery
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Miranda Lam, MD, Radiation Oncologist, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-450
Record Dates: First submitted 2025-01-27; First posted 2025-02-06 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-05

CONDITIONS: Retroperitoneal Sarcoma
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hypofractionated Radiation Therapy (Experimental): This group is receiving hypofractionated radiation therapy (shorter course of radiation therapy)
  Interventions: Radiation: Radiation Therapy; Radiation: Hypofractionationed Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — In this study, patients will receive a hypofractionated course of radiation therapy of 2.85 Gy x 15 fractions (42.75 Gy). If there are 2 or more patients with dose-limiting toxicities, the radiation course will be de-escalated to 2.7 Gy x 15 fractions (40.5 Gy).
Radiation: Hypofractionationed Radiation Therapy — This group is receiving hypofractionated radiation therapy (shorter course of RT)

SUMMARY:
To determine the safety of moderately hypofractionated radiation in the treatment of primary and locally recurrent RPS, based on the evaluation of acute radiation-related toxicity profile of each participant (30-day radiation toxicity)

DETAILED DESCRIPTION:
To determine the safety of moderately hypofractionated radiation in the treatment of primary and locally recurrent RPS, based on the evaluation of acute radiation-related toxicity profile of each participant (30-day radiation toxicity)

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a histologically confirmed STS of the retroperitoneal space or infra-peritoneal spaces of pelvis
* Participant must have radiologically measurable disease (RECIST 1.1), as confirmed by abdomino-pelvic CT or MRI
* Participant must have primary, locally recurrent, or metastatic disease requiring treatment of the retroperitoneal mass
* Tumor must be suitable for radiotherapy and surgery based on pre-treatment CT scan/MRI in multidisciplinary discussion with surgeon and radiation oncologist (anticipated macroscopically complete resection, R0/R1 resection)
* Age: 18 years or older
* ECOG performance status ≤2
* Absence of history of bowel obstruction, mesenteric ischemia, or severe chronic inflammatory bowel disease.
* Normal renal function (calculated creatinine clearance ≥50 mL/min)
* Normal bone marrow and hepatic function (white blood cell count ≥2·5 × 10⁹ cells per L, platelet count ≥80 × 10⁹ cells per L, and total bilirubin <2 times upper limit of normal)
* Women of child-bearing potential must have a negative pregnancy test within 3 weeks prior to the first day of study treatment
* Patients capable of childbearing/reproductive potential should use adequate contraception
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Sarcoma originating from bone structure, abdominal or gynecological viscera
* Any of the following histological subtypes: gastrointestinal stromal tumor, rhabdomyosarcoma, primitive neuroectodermal tumor or other small round blue cell sarcoma, osteosarcoma, chondrosarcoma, aggressive fibromatosis, or sarcomatoid or metastatic carcinoma
* Prior RT to the RPS
* Prior abdominal or pelvic irradiation for other prior malignancy or other disease
* Prior different invasive malignancy may be eligible per the discretion of the treating investigator and review by the Principal Investigator (PI)
* Prior chemotherapy or immunotherapy within 6 weeks of start of RT
* Pregnant women are excluded from this study because RT has the potential for teratogenic or abortifacient effects.
* HIV-positive individuals on combination antiretroviral therapy are ineligible because of the potential for increased sensitivity to RT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Side effects from radiation therapy | From enrollment to 30-days after the completion of radiation treatment
  Evaluation of acute radiation-related toxicity profile of each participant, specifically nausea, vomiting, diarrhea, and other gastrointestinal (GI) side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Miranda Lam, Principal Investigator — Dana-Farber/Brigham and Women's Cancer Center
Locations (1):
- Brigham and Women's Hospital / Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF